CLINICAL TRIAL: NCT05580705
Title: Effects of Vibration Therapy in Addition to Routine Physical Therapy on Pain, Balance, Functional Disability and Satisfaction in Patients With Diabetic Neuropathy
Brief Title: Effects of Vibration Therapy in Addition to Routine Physical Therapy in Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sajawal Bashir
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetes Mellitus; Vibration Therapy; Diabetic Neuropathy; Pain; Balance; Functional Disability; Patient satisfaction; Routine Physical Therapy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Pain; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It will be a single blinded study and the outcome assessor will be blinded to the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROUTINE PHYSICAL THERAPY GROUP (Active Comparator): This group will receive routine physical therapy including strength training intervention. This protocol will be given for two weeks (6 sessions on alternate days, 3 sessions per week), outcomes will be measured at baseline, at the end of 1st week and 2nd week.
  Interventions: Other: Routine Physical Therapy
- VIBRATION THERAPY (Experimental): This group will receive routine physical therapy and vibration therapy. This protocol will be given for two weeks (6 sessions on alternate days, 3 sessions per week), outcomes will be measured at baseline, at the end of 1st week and 2nd week.
  Interventions: Other: Vibration Therapy

INTERVENTIONS:
Other: Routine Physical Therapy — The Routine Physiotherapy treatment will include Transcutaneous Electrical Nerve Stimulation, Hot pack, Range of Motion (ROM) Exercises and Muscle Strengthening Exercises
  Arms: ROUTINE PHYSICAL THERAPY GROUP
Other: Vibration Therapy — Vibration Therapy will include a vibration device of brand Manipol, model number RK-001. It has 360 degree off-centered axis with a frequency of 2500 times per minute. It will be applied on sole of the foot for about 15 mins.
  Arms: VIBRATION THERAPY

SUMMARY:
The study is aimed to determine the effects of sole-foot vibration therapy on pain intensity, static and dynamic balance, functional status and satisfaction to the intervention applied on patients with peripheral neuropathy due to type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Peripheral Diabetic Neuropathy has disastrous effects on human body. It causes impairment which makes normal functioning and activity of daily life difficult. Vibration therapy improves neural mechano-sensitivity to promote movement and function.

In Pakistan, researches have been conducted only on Whole-body vibration and no data is available on foot-sole vibration therapy which is convenient to apply and appropriate for patients as there will be no fear of fall associated during treatment. Therefore, the aim of this study is to analyze the effects of vibration therapy, applied locally on foot, on pain management, balance adjustment, function and satisfaction to treatment in patients with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age of 40-75 years
* Both male and female participants
* On oral medicine for diabetes
* HbA1C <8.5%, and controlled blood sugar in the last three months
* Patients with < 6 years from diagnosis of diabetes
* Diagnosed patient of peripheral neuropathy having type 2 diabetes by registered medical practitioner
* Patient is able to stand on both feet.

Exclusion Criteria:

* Systemic diseases such as advanced cardiovascular, renal, or hepatic diseases
* Open wounds/ulcers on lower limb
* Neurological illness that affects balance i.e. vertebral artery syndrome, Multiple Sclerosis, Parkinson's disease, Alzheimer's disease, Stroke and cerebral ataxia
* Musculoskeletal problems such as leg length discrepancy, ankle sprain and severe osteoarthritis of knee and hip joints
* Patients who have performed vibration therapy exercises prior to intervention
* Patient under any antihypertensive drugs and blood pressure more than 160/95 mm hg

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Change in pain score will be measured at baseline, at the end of 1st week and 2nd week.
  Pain Intensity will be measured by using Numeric Pain Rating Scale. Pain score range from 1-10, with 1 indicates least possible pain level and 10 is the worst pain level.
Dynamic and Static Balance | Change in Balance score will be measured at baseline, at the end of 1st week and 2nd week.
  Dynamic and static balance will be measured by using Berg Balance Scale. Its score range from 0 to 56, lower score represents more chances of losing balance and requirement of assistive measures.
Level of Functional Disability | Change in Functional Disability score will be measured at baseline, at the end of 1st week and 2nd week
  Functional Disability will be measured by using Revised Neuropathy Disability Score. The total score is 10 with higher score indicates more severity of disease.
Patient Satisfaction Level | Change in Patient Satisfaction Level will be measured at baseline, at the end of 1st week and 2nd week.
  Patient Satisfaction Level will be measured by the Patient Satisfaction Questionnaire. Total score is 90. and higher score towards maximum value indicates higher level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Immediately after publication
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending on 36th month

REFERENCES:
- [Derived] Bashir S, Jamil A, Ali S. Effects of vibration therapy with routine physical therapy on pain, balance, and functional disability in diabetic neuropathy patients: a randomised controlled trial. J Pak Med Assoc. 2025 Apr;75(4):534-539. doi: 10.47391/JPMA.20058. PMID 40269358